CLINICAL TRIAL: NCT06984705
Title: Epidemiological and Clinical Characteristics of Human Mpox Outbreak in Equateur Province in the Democratic Republic of Congo (Part3)
Status: Enrolling by invitation | Type: Observational
Sponsor: Osaka Metropolitan University (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Principal Investigator, Natsuko Kaku, Lecturer, Osaka Metropolitan University
Other Study IDs: N553/BN/PMMF/2024-3
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Mpox (Monkeypox)
Keywords: vaccine efficacy; test negative control
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin lesion and oral mucosa swab sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- cases: • Cases are defined as Individuals who reported to local health agents with symptoms consistent with mpox and subsequently tested positive for mpox through a molecular-based diagnostic test.
- controls: Controls are defined as Individuals who reported to local health agents with symptoms consistent with mpox but subsequently tested negative for mpox through a molecular-based diagnostic test.

SUMMARY:
The goal of this study is to evaluate the effectiveness of smallpox vaccination administered before the global eradication of smallpox against currently circulating mpox in the Democratic Republic of the Congo.

The main question it aims to answer is:

Is the smallpox vaccine experience protective against mpox infection ?

Researchers will compare mpox test positive group and negative group to see if the smallpox vaccine can protect against mpox infection.

Participants will

* be included after informed consent,
* respond the survey with structured questionnaire
* and accept skin lesion and blood sampling.

DETAILED DESCRIPTION:
Mpox is caused by the monkeypox virus (MPXV), a member of the genus Orthopoxvirus (family Poxviridae). This virus is closely related to the variola virus, which causes smallpox. MPXV was first identified in 1958, and the first human case was reported in Democratic Republic of the Congo (DRC) in 1970. It was presumed that the smallpox vaccine would confer cross-protection against mpox. Following the global eradication of smallpox in 1980, mpox remained largely confined to limited regions in Central Africa-where zoonotic spillover from wild animal reservoirs constituted the primary route of transmission. Equateur Province is among the areas in the DRC with a notably high burden of reported mpox cases.

Over the past five decades, routine smallpox vaccination ceased worldwide, resulting in waning herd immunity against orthopoxviruses. During this period, mpox incidence rose markedly, with an estimated tenfold increase in global cases. Two principal genetic clades of MPXV have been identified: clade I (historically referred to as the Congo Basin clade) and clade II (the West African clade). In 2018, Nigeria experienced a resurgence of mpox, highlighting the virus's potential to emerge in previously controlled areas. Starting in 2022, clade II mpox circulated globally, especially among men who have sex with men (MSM), peaking in mid-2022 before declining to persistently lower levels by early 2023. Although clade II mpox typically exhibits a low case-fatality ratio (<1%), clade I has historically been associated with more severe disease and higher mortality. In 2023, the number of reported mpox cases continued to climb in the DRC, prompting the World Health Organization (WHO) to declare a Public Health Emergency of International Concern (PHEIC) in August 2024.

Recent surveillance indicates that sub-clade Ia MPXV is spreading in western DRC through multiple transmission modes, including contact with infected wild animals, household exposure, or sexual contact. By contrast, sub-clade Ib mpox in the eastern part of the country appears initially to spread via intimate or sexual contact between adults, followed by household transmission. Numerous environmental and social risk factors-including the consumption of rodent species, deforestation, climate change, civil unrest, population displacement, emerging MPXV variants, and weakened immunity-may be driving mpox incidence. Clade Ia mpox is currently affecting western parts of the DRC, yet the epidemiology remains poorly understood due to the limited number of laboratory-confirmed cases.

This study aims to characterize the clinical features of the 2024 mpox outbreak in Equateur Province of DRC and to identify associated risk factors. The findings will advance understanding of mpox transmission dynamics and disease severity, ultimately informing more effective prevention and control strategies in endemic settings.

The overall aim of this study is to describe the clinical characteristics of the 2024 mpox outbreak in the DRC and to identify associated risk factors. This research comprises three components: 1) a case-control study, 2) a transmission study, and 3) a vaccine effectiveness study.

And this protocol is for 3) a vaccine effectiveness study aim to evaluate the effectiveness of smallpox vaccination administered before the global eradication of smallpox against currently circulating mpox.

ELIGIBILITY:
Inclusion Criteria:

* Individuals born before 1984: Although it is officially stated that smallpox vaccination was administered in the DRC until 1982, individuals born up to 1984 were included to account for potential discrepancies of several years in remote areas.
* Presence of skin lesions suspected to be mpox.
* Provision of informed consent:

Proxy-assisted informed consent is allowed under safety considerations. Following oral consent, the investigator will document this on the informed consent form as a witness.

Exclusion Criteria:

Participants will be excluded from the study under the following conditions:

• Refusal to participate in the study: Individuals who decline to provide consent for study participation will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study targets patients born before 1984 with mpox-like skin lesions (both sexes) in the selected sites. All patients suspected of having mpox-like lesions and who provide proxy-assisted written informed consent to participate in the study are eligible for inclusion due to reduction of the risk of contact transmission with verbal agreement documented and confirmed by a witness. This approach prioritizes participant and staff safety while adhering to ethical standards.
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Confirmed mpox | Day 1
  Definition: the positivity of mpox is determined based on the gene amplification testing for mpox genes.
  The subjects sampled as suspected mpox patients will be classified based on pathogen diagnostic results: those testing positive will be defined as cases, and those testing negative will be defined as controls.

SECONDARY OUTCOMES:
Severity | Day 1
  Mpox severity will be evaluated based on skin lesion burden, clinical complications, organ dysfunction, and mortality outcomes.
  Scoring Criteria:
  Mild: Fewer than 25 lesions. Moderate: 26-99 lesions. Severe: 100 or more lesions or the presence of organ dysfunction, regardless of lesion count.
  Fatal Outcome: If a patient dies from mpox or its complications during the study, the case will be classified as "fatal outcome." Assessment: The severity score will integrate the number of skin lesions across various anatomical sites and documented signs of complications (e.g., respiratory distress, neurological symptoms, renal impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Natsuko Kaku, PhD, Principal Investigator — Osaka Metropolitan University
Locations (1):
- Equateur Provincial Public Health Laboratory, Mbandaka, Équateur Province, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided